CLINICAL TRIAL: NCT05134714
Title: "Evaluation of Clinical Performance and Success Rate of CAD/CAM Versus Conventional Band and Loop Space Maintainer Randomized Clinical Trial and in Vitro Study"
Brief Title: "Evaluation of Clinical Performance and Success Rate of CAD/CAM Versus Conventional Band and Loop Space Maintainer"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, sara Abdelkhalek hassan younes, assistant teacher, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PED 21-4D
Record Dates: First submitted 2021-11-02; First posted 2021-11-26 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: CAD/CAM Space Maintainer
Keywords: space maintainer; CAD/CAM space maintainer

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1(study group): CAD/CAM zircon band and loop space maintainer (Experimental): Solid monolithic zirconia material which utilizes CAD/CAM technology for its designing and milling of the restoration will be used for fabrication of the space maintainer.
  Interventions: Device: CAD/CAM zircon band and loop space maintainer; Device: Conventional metal band and loop space maintainer
- Group 2(control): Conventional metal band and loop space maintainer (Active Comparator): Stainless steel band and loop space maintainer will be made. Stainless steel appropriate band will be selected according to the size of the abutment teeth then design of the loop will be obtained, then will be send to the laboratory for soldering.
  Interventions: Device: CAD/CAM zircon band and loop space maintainer; Device: Conventional metal band and loop space maintainer

INTERVENTIONS:
Device: CAD/CAM zircon band and loop space maintainer — Solid monolithic zirconia material which utilizes CAD/CAM technology for its designing and milling of the restoration will be used for fabrication of the space maintainer.
  Other Names: CAD/CAM space maintainer
Device: Conventional metal band and loop space maintainer — Stainless steel appropriate band will be selected according to the size of the abutment teeth and then design of the loop will be obtained, then will be send to the laboratory for soldering.
  Other Names: metal band and loop space maintainer

SUMMARY:
This study is to evaluate and compare CAD/CAM zircon space maintainer and conventional metal of band and loop space maintainers in terms of plaque deposits and gingival health and, the success rate of the appliances in terms of: survival time, cement loss and appliance breakage. And to compare both appliances in terms of patient satisfaction.

This study consists of two parts: in vivo part (split mouth RCT) and in vitro part:

In vivo study:

Its sample size was found to be (36) cases (i.e. 18 case per group). Sample size calculation was performed using G*Power version 3.1.9.7 Sample size will be increased by about 10% to compensate for the drop-out.

In this in vivo study split mouth will be randomly divided into two groups:

Group 1: Conventional metal band and loop space maintainer Group 2: CAD/CAM zircon band and loop space maintainer

In vitro study:

its sample size was found to be (24) samples (i.e. 8 samples per group). Sample size calculation was performed using G*Power version 3.1.9.7 Sample size will be increased by about 10% to compensate for the drop-out.

Grouping:

The zirconia specimen divided randomly into three groups according to type of cements:

Group 1: Self-adhesive resin cement Group 2: Resin-modified glass ionomer cement Group 3: Universal bioactive cement

DETAILED DESCRIPTION:
Introduction:

Primary teeth play an important role in the development and growth of a child. Although their role in esthetics, speech, eating, and to encourage normal function. The other main function of a primary tooth is to hold space for the permanent successor until it's time for eruption. This normal physiologic process can be affected due to early premature loss of primary molars, due to dental caries which may lead to mesial tipping or migration of large permanent molar teeth into the space created. This may result in loss of space leading to discrepancy of arch length, malocclusion, crowding of teeth, cross bite, impaction of permanent premolars, and supra-eruption of opposing tooth. The best approach to maintain arch space and to prevent malocclusion is to use a space maintainer. Band and loop has been used since long as a space maintainer with high success rates. But there are some disadvantages can be associated with space maintainers which include, loss of cement, solder failure, caries formation along the margins of the band, long construction time, and the possibility of metal allergy in some patients. These shortcomings in addition to the rising interest of esthetic dentistry augmented by advances in technology have led to the development of newer materials and designs in the fabrication of space maintainers such as fiber-reinforced composite resins (FRCR) as fixed space maintainers. Digital technologies such as CAD CAM technology and new materials are becoming popular, getting better and changing the way to therapy. The ceramic space maintainer seems to be a suitable alternative to the conventional band and loop space maintainer. The appliance is well tolerated by the patient and also gives the benefit of advanced aesthetics with improved strength and allowing the easiest way of debonding during eruption of permanent successors.

The aim of the current study is:

A) Primary Objective Evaluate and compare CAD/CAM zircon space maintainer and conventional metal of band and loop space maintainers in terms of plaque deposits (Plaque index), gingival health (Gingival index).

The success rate of appliances in terms of survival time, cement loss and appliance breakage.

B) Secondary Objectives Compare both appliances in terms of patient satisfaction. Evaluate the shear bond strength of three different cements used for CAD CAM zircon space maintainer cementation in vitro.

This study consists of two parts: in vivo part (split mouth RCT) and in vitro part:

1- In vivo study:

Study design:

A split mouth Randomized controlled clinical trial (RCT)

In this in vivo study split mouth will be randomly divided into two groups:

Group 1(study group): CAD/CAM zircon band and loop space maintainer Group 2(control): Conventional metal band and loop space maintainer Interventions

All interventions will be performed by the primary investigator as follows:

Control group:

1. Stainless steel appropriate band will be selected according to the size of the abutment teeth.
2. Then the band will be seated on the tooth and full arch impression will be obtained using alginate material.
3. The band will be removed gently and then stabilize in the impression material.
4. Maxillary impression will be obtained using alginate material.
5. Impressions will be poured in stones and then design of the loop will be obtained, then will be send to the laboratory for soldering.
6. Afterwards abutment teeth will be cleaned.
7. Isolations precautions will be taken.
8. Cementing the space maintainer using glass ionomer cement.
9. Any excess material will be removed. Study group

1. Impression of the upper and lower arches will be taken using elastomeric impression material.

2. Impressions will be send to the lab for fabrication of zircon space maintainer.

3. Solid monolithic zirconia material which utilizes CAD/CAM technology for its designing and milling of the restoration will be used for fabrication of the space maintainer.

4. Lab Procedure: zircon CAD/CAM-fabricated material has to be digitally designed by a technician using a digital scanner and design software.

5. CAD CAM space maintainer will be cemented. Oral hygiene instructions will be given to patients as a standard of care after dental procedures.

Clinical evaluation Clinical evaluation of success rates of the modalities regarding survival time, cement loss, breakage of the appliances.

Plaque index, that is running in a scale from 0 to 3 where 0 means no plaque,1 film of plaque adhering to free gingival margin,2 moderate accumulation of soft deposits on the tooth and gingival margin, and 3 means abundance of soft debris (according to the PI described by Silness & Loe) Gingival health, scores from 0 to 3 where 0 no inflammation, 1slight redness no bleeding on probing, 2 redness and bleeding on probing, and 3 severe inflammation with edema and ulceration to spontaneous bleeding (according to the GI described by Silness & Loe), and patient satisfaction (checked using visual analogue scale (six point facial Wong-Baker Scale) in vivo.

Follow up and outcome:

Patients will be recalled for clinical follow up after 3, 6, 9 and 12 months. 2- In vitro study:

Materials:

Three different cements, namely, self-adhesive resin cement, resin-modified glass ionomer cement, and universal bioactive cement, will be used in this study. All of the materials will be applied according to the manufacturers' instructions.

Grouping:

The zirconia specimen divided randomly into three groups according to type of cements:

Group A: Self-adhesive resin cement Group B: Resin-modified glass ionomer cement Group C: Universal bioactive cement

Specimen collection and Preparation for shear bond strength:

Freshly extracted human molars, caries free will be collected and examined by stereomicroscope to exclude any specimen with cracks.

The roots of each tooth will be removed, the teeth will be cleaned and polished with non-fluoridated flour of pumice for 10s using rubber cup, and then rinsed with stream of water and then drying it.

Teeth will be mounted in a self-cure acrylic resin so that the crown will be exposed, the acrylic blocks will be number coded with a different number for each group of samples.

Preparation of zirconia specimens Zirconia specimens will be milled from yttrium-stabilized tetragonal zirconia (Y-TZP). The bonding site of each specimen will be finished using 600-, 800-, 1000- and 1200-grit silicon carbide paper to obtain a flat surface. All the zirconia specimen will be ultrasonically cleaned in deionized water for 5 min and divided into three groups according to the types of cements.

Cementation protocol The zirconia specimens will be divided into three groups according to type of cement.

The zirconia specimens will be bonded to the enamel specimen of the extracted teeth by cement prepared according to the manufacturer's instructions. Excess cement was removed.

Specimens will be held in a fixed position without any movement for 5 min to achieve self-curing without motion.

Shear Bond Strength testing After the cementation procedure, all specimens will be stored at 37°C in distilled water for 24 h. Then, the specimens will be subjected to Shear Bond Strength testing by applying a shear load to the zirconia until bond failure occurred.

Following deboning, the specimen will be examined under a stereomicroscope to determine the mode of bond failures (adhesive, cohesive, or mixed).

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged :

   A-minimum:4years B-maximum: 7 years old
2. Patients who are medically free
3. Premature loss of bilateral primary molar.
4. Sound and healthy buccal and lingual surfaces of selected primary molars.

Exclusion Criteria:

1. Children with dental abnormalities (cross bite, open bite, and deep bite).
2. Parafunctional oral habits.
3. Carious lingual and buccal surfaces of primary molars.
4. Lack of patient/parent compliance and cooperation.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical success: Evaluate and compare CAD/CAM zircon space maintainer and conventional metal of band and loop space maintainers in terms of plaque deposits (Plaque index) | Up to 12 months
  Plaque index, that is running in a scale from 0 to 3 where 0 means no plaque,1 film of plaque adhering to free gingival margin,2 moderate accumulation of soft deposits on the tooth and gingival margin, and 3 means abundance of soft debris.
Clinical success: Evaluate and compare CAD/CAM zircon space maintainer and conventional metal of band and loop space maintainers in terms of Gingival health, by assessing the gingival index. | up to 12 months
  Gingival health, scores from 0 to 3 where 0 no inflammation, 1slight redness no bleeding on probing, 2 redness and bleeding on probing, and 3 severe inflammation with edema and ulceration to spontaneous bleeding,47 and patient satisfaction.
The success rate of appliances in terms of survival time. | Up to 12 months
  Clinical evaluation of success rates of the modalities regarding survival time by checking both space maintainers and identify if there is cement loss or breakage of the appliances during the follow up period.

SECONDARY OUTCOMES:
Compare both appliances in terms of patient satisfaction. | Up to 12 months
  patient satisfaction by (checked using visual analogue scale )patients will be choose from smiley faces if they are happy or not

CONTACTS AND LOCATIONS:
Overall Officials: Gehan G. Allam, PHD, Study Chair — Ain Shams Univesity

IPD SHARING:
Plan to Share IPD: No